CLINICAL TRIAL: NCT02507583
Title: Phase I Study in Humans Evaluating the Safety of Rectus Sheath Implantation of Diffusion Chambers Encapsulating Autologous Malignant Glioma Cells Treated With Insulin-like Growth Factor Receptor-1 Antisense Oligodeoxynucleotide (IGF-1R/AS ODN) in 32 Patients With Newly Diagnosed Malignant Glioma
Brief Title: Antisense102: Pilot Immunotherapy for Newly Diagnosed Malignant Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: david andrews (Other)
Responsible Party: Sponsor-Investigator, david andrews, Chief, Division of Neuro-Oncology, Thomas Jefferson University
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14G.96; JT 5979 (Other: JeffTrial Number)
Record Dates: First submitted 2015-06-29; First posted 2015-07-24 (Estimated); Last update posted 2025-05-07 (Actual); Status verified 2020-10

CONDITIONS: Malignant Glioma; Neoplasms
Keywords: Brain Tumor; Glioma; Newly Diagnosed
MeSH Terms: conditions — Glioma; Neoplasms; Brain Neoplasms | interventions — Surgical Procedures, Operative; Tissue and Organ Harvesting; Craniotomy; Drug Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cohort 1 (Experimental): After protocol amendment dated 11 May 2017, all subjects enrolled into the trial will receive 20 chambers for 48 hours.
  Interventions: Drug: IGF-1R/AS ODN; Surgery with tissue harvest and implantation 20 diffusion chambers in the rectus sheath with IGF-1R/AS ODN within 24 hours of craniotomy, implanted for 48 hours.

INTERVENTIONS:
Drug: IGF-1R/AS ODN; Surgery with tissue harvest and implantation 20 diffusion chambers in the rectus sheath with IGF-1R/AS ODN within 24 hours of craniotomy, implanted for 48 hours.
  Other Names: Insulin-like growth factor receptor-1 antisense oligodeoxynucleotide

SUMMARY:
This human Phase 1 trial is a continuation of a Phase 1 trial which enrolled patients with recurrent gliomas (#TJU-14379-101) and which was designed after a previously conducted Phase 1 human trial at our institution. With certain modifications, it is intended to reproduce the safety results of the recurrent glioma previous trials as well as explore any objective clinical responses in newly diagnosed patients. Protocol 14379-101 is closed to accrual and Abbreviated Clinical Report is prepared for FDA submission. The safety profile for this protocol was quite favorable.

This treatment involves taking the patient's own tumor cells at surgery, treating them with an investigational new drug (an antisense molecule) designed to shut down a targeted surface receptor protein, and re-implanting the cells, now encapsulated in small diffusion chambers the size of a nickel in the patient's abdomen within 24 hours after the surgery. Loss of the surface receptor causes the tumor cells to die in a process called apoptosis. As the tumor cells die, they release small particles called exosomes, each full of tumor antigens. The investigators believe that these exosomes as well as the presence of the antisense molecule work together to activate the immune system against the tumor as they slowly diffuse out of the chamber. Immune cells are immediately available for activation outside of the chamber because a wound was created to implant these tumor cells and a foreign body (the chamber) is present in the wound. In this trial, a dose escalation of the therapeutic agent will involve an increase in both biodiffusion chamber number as well as the time the biodiffusion chambers remain implanted. The wound and the chamber fortify the initial immune response which eventually leads to the activation of immune system T cells that attack and eliminate the tumor. By training the immune system to recognize the tumor, the patient is also protected through immune surveillance from later tumor growth should the tumor recur. Compared to treatment alternatives for tumor recurrence, including a boost of further radiation and more chemotherapy, this treatment represents potentially greater benefit with fewer risks.

DETAILED DESCRIPTION:
This trial will be an adaptation of Protocol 101 which recently closed after rapid and complete accrual, now with an escalation of the induction vaccination in four cohorts. For practical purposes, a standard dose-escalation study is not possible with the current paradigm. Although the investigators may have identified a distinct bioactive byproduct of Insulin-like growth factor receptor-1 Antisense Oligodeoxynucleotide (IGF-1R/AS ODN)-induced tumor cell apoptosis (exosomes), it is difficult to perform a dose escalation in a typical fashion. Also, antigen concentration can affect immune response in a biphasic manner: too little or too much can dampen an immune response, so even if the antigen or antigens were known, a typical pharmacologic dose escalation would not follow typical pharmacokinetics. For these reasons, in Protocol 102, 32 patients will have therapy at initial surgery followed by implantation of 20 chambers for a duration of 48 hours. There was a documented increase in tumor infiltrating lymphocytes after treatment in our original trial, this observation provided preliminary supporting evidence that this therapeutic vaccine will elicit an adaptive immune response. Protocol 102 has been designed to further elucidate an immune response with a quantitative assessment of tumor specific T cells as well as circulating M2 macrophages before and after treatment. The design of the Phase 1 trial will allow a statistical analysis of both antigen dose (number of chambers) and time of exposure (chamber dwell time) as either variable may relate to any toxicity or treatment response.

A summary of the treatment paradigm includes: Pre-operative plasma leukopheresis, then surgery with tissue harvest and implantation of 20 diffusion chambers in the rectus sheath with IGF-1R/AS ODN as previously reported within 24 hours of craniotomy, implanted for 48 hours. All patients who meet the eligibility criteria and agree to participate in this study will be potential candidates for therapy.

ELIGIBILITY:
Inclusion Criteria:

* Documentation by MR of a gadolinium-enhancing intraparenchymal mass consistent with malignant glioma.
* Frozen section diagnosis of WHO Grade IV glioma, confirmed with permanent section and immunopositive for IGF-1R.
* An Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2 or a Karnofsky Performance Score (KPS) of at least 60.
* Must be 18 years of age or older.
* Must sign an approved informed consent.
* Hemodynamically stable, consistent with Standard of Care values for patients undergoing elective tumor resection.

Exclusion Criteria:

* Females who are pregnant, nursing, or not inclined to use adequate contraceptive methods if necessary to prevent pregnancy during the study.
* An active second primary malignancy with the exception of basal cell or squamous cell skin carcinoma.
* Major concomitant medical illness inclusive of severe chronic obstructive pulmonary disease, multiple sclerosis, symptomatic coronary artery disease, heart failure, recent major cerebrovascular accident, brittle diabetes, renal dialysis, end stage liver disease, labile hypertension, or any autoimmune disorder.
* A history of heparin-induced thrombocytopenia or hypersensitivity to heparin, enoxaparin, or pork products.
* An abnormal International Normalized Ratio (INR) of greater than 1.3, if repeatable and refractory to correction by routine methods.
* Documented deep venous thrombosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2018-03-06 (Actual); Study Completion 2020-08-17 (Actual)

PRIMARY OUTCOMES:
Collect adverse events as a measure of safety and tolerability of IG-1R/ AS ODN | 36 months
  Adverse events and survival outcomes will be captured as a measure of safety and tolerability of IG-1R/AS ODN administered as a treatment 4 to 6 weeks before initiation of standard of care treatment. Blood (equivalent of 8 units of mononuclear cells by plasma leukopheresis) will be collected within 3 days of craniotomy and 7 tbsp of blood on days 14, 28, 42, 56, followed by every 3 months after vaccination to measure the degree of anti-glioma Cytotoxic T lymphoctye immunity achieved.

SECONDARY OUTCOMES:
Document any T-1 weighted MRI-based radiographic responses to treatment. | Evaluated 3 days pre surgery, and again at day 28, day 56, and then every 3 months up to 24 months.
  T-1 weighted abnormalities include: (1) size of the enhancing area utilizing the broadest unambiguous diameter in any orthogonal plane; (2) characteristics of the enhancement (e.g. progression from linearity to nodularity or regression from nodularity to linearity) and (3) intensity of enhancing area
Document any T-2 weighted MRI-based radiographic abnormalities or responses to treatment. | Evaluated 3 days pre surgery, and again at day 28, day 56, and then every 3 months up to 24 months.
  T-2 weighted abnormalities include: (1) local mass effect; (2) size of T-2 weighted abnormality (e.g. edema, tumor, radiation change); (3) invasion of the deep white matter tracts; and (4) distal progression.
MRI measure of tumor response | Evaluated 3 days pre surgery, and again at day 28, day 56, and then every 3 months up to 24 months.
  Each imaging characteristic will be rated as increased, decreased, or without change. Since distal progression including invasion of the contralateral hemisphere will either be present or absent, this criterion will be scored as either absent (stable) or present utilizing FLAIR sequence. Comparisons will be made between an MRI study performed within 48 hours of craniotomy documenting residual contrast-enhancing tumor.

OTHER OUTCOMES:
Measurement of Immune response | 36 months
  After the treatment, serial measurements of cytokines, chemokines, and peripheral blood mononuclear cells will be performed from obtained blood samples as outcome measurements of immune response.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Judy, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Andrews DW, Resnicoff M, Flanders AE, Kenyon L, Curtis M, Merli G, Baserga R, Iliakis G, Aiken RD. Results of a pilot study involving the use of an antisense oligodeoxynucleotide directed against the insulin-like growth factor type I receptor in malignant astrocytomas. J Clin Oncol. 2001 Apr 15;19(8):2189-200. doi: 10.1200/JCO.2001.19.8.2189. PMID 11304771
- [Derived] Andrews DW, Judy KD, Scott CB, Garcia S, Harshyne LA, Kenyon L, Talekar K, Flanders A, Atsina KB, Kim L, Martinez N, Shi W, Werner-Wasik M, Liu H, Prosniak M, Curtis M, Kean R, Ye DY, Bongiorno E, Sauma S, Exley MA, Pigott K, Hooper DC. Phase Ib Clinical Trial of IGV-001 for Patients with Newly Diagnosed Glioblastoma. Clin Cancer Res. 2021 Apr 1;27(7):1912-1922. doi: 10.1158/1078-0432.CCR-20-3805. Epub 2021 Jan 26. PMID 33500356